CLINICAL TRIAL: NCT05967468
Title: Evaluation of Family-Based Behavioral Treatments for Youth With Anxiety and Obsessive-Compulsive Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Eric A Storch, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-53969
Record Dates: First submitted 2023-07-12; First posted 2023-08-01 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Obsessive-Compulsive Disorder in Children; Anxiety Disorder of Childhood; Social Anxiety Disorder of Childhood; Obsessive-Compulsive Disorder in Adolescence; Generalized Anxiety Disorder; Separation Anxiety; Panic Disorder; Panic Disorder With Agoraphobia; Panic Attacks
Keywords: obsessive-compulsive disorder; anxiety; cognitive-behavioral therapy; children
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety, Separation; Panic Disorder; Obsessive-Compulsive Disorder; Anxiety Disorders | interventions — Bibliotherapy

STUDY DESIGN:
Intervention Model Description: Children (N=100), ages 7-13 will be randomized to one of three conditions
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor is blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Family-Based Internet-Based CBT Group (iCBT) (Experimental): One third of participants will be randomized to receive iCBT. Each week of treatment, the parent will be encouraged to read the corresponding materials on the Baylor College of Medicine (BCM) webpage, complete accompanying worksheets, and guide their child through completing activities in the child-facing materials, with support from a therapist (6 30-minute supportive videoconferencing via Zoom, 6 emails on alternating weeks). One core aspect of treatment will be parents leading their child through graduated exposure. Exposures, a hallmark of CBT for anxiety, are used to gradually and repeatedly confront feared stimuli. For example, exposure therapy for a child fearful of dogs may begin with looking at pictures of dogs and standing across the park from a dog on a leash, to eventually petting a dog. All relevant information regarding parent-led exposures will be detailed in the treatment materials, and therapists will review with parents via email and/or video-conferencing sessions.
  Interventions: Behavioral: Family Based, Internet-Based Cognitive Behavioral Therapy
- Parent Training Bibliotherapy (SPACE) (Experimental): One third of participants will be randomized to the SPACE group. Families will receive 4 45-minute supportive video calls with a therapist over the course of 12-14 weeks. Participating families will receive a copy of the book 'Breaking Free of Child Anxiety and OCD' to use at home and in session with the therapist. During each of the video-conferencing sessions, therapists will serve to provide encouragement and support as the parent works through the program independently.
  Interventions: Behavioral: Bibliotherapy, low therapist contact SPACE
- Active Comparator (Active Comparator): One third of participants will be randomized to receive a Relaxation and Mentorship. This involves attending 4 45-minute sessions with a therapist over the course of 12-14 weeks. Topics covered include breathing slowly and deeply, coloring activities, and releasing muscle tension to reduce stress levels.
  Interventions: Other: Relaxation and Mentorship

INTERVENTIONS:
Behavioral: Family Based, Internet-Based Cognitive Behavioral Therapy — Family-based cognitive behavioral therapy employing internet-delivered modules and videos
  Arms: Family-Based Internet-Based CBT Group (iCBT)
Behavioral: Bibliotherapy, low therapist contact SPACE — Parent-based bibliotherapy for treating anxiety disorders in youth
  Arms: Parent Training Bibliotherapy (SPACE)
Other: Relaxation and Mentorship — Relaxation based treatment
  Arms: Active Comparator

SUMMARY:
Anxiety and obsessive-compulsive disorders are among the most common in children. Although cognitive behavioral therapy (CBT) is an effective and evidence-based treatment for such disorders, access to CBT is often limited. Family-based and internet-delivered therapy is one method to increase access to care. The purpose of this project is to evaluate the comparative efficacy and treatment mechanisms of two lower-intensity but effective treatments for families of children with anxiety or obsessive compulsive disorder (OCD) via telehealth compared to an adapted Relaxation and Mentorship Training (RMT) intervention involving breathing exercises with a therapist.

DETAILED DESCRIPTION:
Cognitive-behavioral therapy (CBT) is an effective treatment for anxiety, yet access to CBT is limited for most families due to the cost, practicalities of attending in-person treatment sessions, and limited availability of trained therapists. Low-intensity telehealth delivery of services is a promising method to improve access to care for youth with anxiety and their families, givens its reachability to a wider range of areas (e.g., rural/underserved) and its ability to minimize practical barriers (e.g., treatment could be delivered to home without need for travel), and reduce stigma (e.g., parents do not need to visit mental health clinics). Additionally, parent-involved treatments for youth anxiety are effective and have the potential to reach more children and adolescents who refuse to see a therapist. However, these interventions have not been widely evaluated. The goal of this project is to evaluate the comparative efficacy and treatment mechanisms of two lower-intensity but effective treatments for families of children with anxiety or obsessive compulsive disorder (OCD) via telehealth compared to an adapted Relaxation and Mentorship Training (RMT) intervention involving breathing exercises with a therapist. This study involves two CBT-based intervention groups, both of which have demonstrated efficacy in prior work: 1) a parent-led, therapist-supported Internet based CBT intervention (iCBT) and 2) parent training paired with bibliotherapy intervention (SPACE).

ELIGIBILITY:
Inclusion Criteria:

* The child is between the ages of 7 to 13 years inclusion at enrollment
* The child has clinically significant symptoms of anxiety and/or OCD, as indicated by a score of 12 or higher on the Pediatric Anxiety Rating Scale (PARS).
* The child is appropriate for anxiety-focused treatment (e.g., anxiety is the primary or co-primary problem as diagnosed using the Mini-International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).
* One parent/guardian is able and willing to participate in assessment and treatment (e.g., has sufficient English fluency, the decisional capacity to participate, and can commit to treatment duration).
* The participating parent/guardian lives with their child at least 50% of the time per self-report.
* Both parent and child are able to read and understand English.
* The child has the intellectual and communication skills to engage in CBT, as judged by an experienced supervising clinician.
* Participants must be in the state of Texas for treatment sessions/assessments.

Exclusion Criteria:

* the child has a diagnosis of child lifetime bipolar disorder, drug or alcohol dependence, psychotic disorder, or conduct disorder.
* the child has severe, current suicidal/homicidal ideation and/or self-injury requiring medical intervention (referrals will be made for appropriate clinical intervention).
* the child is receiving concurrent therapy for anxiety.
* New Treatments: Initiation of an antidepressant within 12 weeks before study enrollment OR 6 weeks for an antipsychotic, benzodiazepine, or attention deficit hyperactivity disorder (ADHD) medication before study enrollment. Established Treatment changes: Any change in established psychotropic medication (e.g., antidepressants, anxiolytics, antipsychotic) within 4 weeks before study enrollment. Any medications must remain stable during treatment; downward adjustments due to side effects may be acceptable.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in clinician-rated child anxiety severity throughout the past week. | baseline (before treatment), during treatment (on average 14 weeks), post-treatment (last week of treatment), 1 month follow up
  Each item is scored on a 0 to 5 scale (higher scores correspond to greater severity), yielding a total between 0 and 30.

SECONDARY OUTCOMES:
Anxiety Disorders Interview Schedule (ADIS-IV) with Clinical Severity Ratings | baseline (before treatment), during treatment (on average 14 weeks), post-treatment (last week of treatment), 1 month follow up
  Clinician-rated diagnostic interview that includes current anxiety disorders, depression, obsessive-compulsive disorder, and related disorders. Each diagnostic category is coded as present or absent based on symptom criteria and clinical severity ratings (CSRs), which indicate the level of clinical interference. CSRs are scored on a 0-8 scale (0 = not at all; 8 = very, very much). CSRs of 4 or above indicate the clinical levels.
Clinical Global Impression-Severity | baseline (before treatment), during treatment (on average 14 weeks), post-treatment (last week of treatment), 1 month follow up
  Clinician-rated child psychopathology severity rating. A single item is scored 0-6 (0= no illness; 6= extremely severe symptoms).

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No